CLINICAL TRIAL: NCT03614078
Title: A Phase 2a Study to Evaluate Safety, Tolerability, and Efficacy of PRCL-02 in Patients With Moderate to Severe Chronic Plaque Psoriasis
Brief Title: A Study of PRCL-02 in Moderate to Severe Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: PRCL Research Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRCL-PoC
Record Dates: First submitted 2018-07-30; First posted 2018-08-03 (Actual); Results first posted 2020-03-30 (Actual); Last update posted 2020-03-30 (Actual); Status verified 2020-03

CONDITIONS: Psoriasis Vulgaris; Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- PRCL-02 Dose 1 (Experimental): Loading dose followed by a once daily maintenance dose commencing on Day 2 and continuing for 12 weeks
  Interventions: Drug: PRCL-02
- PRCL-02 Dose 2 (Experimental): Loading dose followed by a once daily maintenance dose commencing on Day 2 and continuing for 12 weeks
  Interventions: Drug: PRCL-02
- Placebo (Placebo Comparator): Loading dose followed by a once daily maintenance dose at matching treatment levels, commencing on Day 2 and continuing for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PRCL-02 — Oral tablets
  Arms: PRCL-02 Dose 1; PRCL-02 Dose 2
Drug: Placebo — Oral tablets
  Arms: Placebo

SUMMARY:
The aim of this study is to evaluate safety, tolerability, and efficacy of PRCL-02 in moderate to severe chronic plaque psoriasis

ELIGIBILITY:
Inclusion Criteria:

* Presents with moderate to severe psoriasis vulgaris based on:

  * Chronic psoriasis vulgaris for at least 6 months
  * Plaque psoriasis involving at least 10% body surface area (BSA)
  * Psoriasis Area and Severity Index (PASI) total score of at least 12
* Have at least 2 evaluable plaques located in 2 different body regions. (Also for participants who elect to have plaques biopsied, should be suitable for a total of 4 punch biopsies each, and one lesion, preferably on a region of the body that is not normally exposed (e.g., trunk), should be selected for biopsy)
* Have a Static Physician's Global Assessment (sPGA) score of greater than or equal to (≥)3
* Are candidates for systemic therapy
* Have a body mass index (BMI) within the range of 18 to 40 kilograms per square meter (kg/m2)
* Women who are of childbearing potential must agree to use 1 highly effective method of contraception, or a combination of 2 effective methods of contraception for the entirety of the study
* Women of non childbearing potential are defined as women who are:

  * Infertile due to surgical sterilization (hysterectomy, bilateral oophorectomy, or tubal ligation), congenital anomaly such as mullerian agenesis; or
  * Post-menopausal, defined as either:

    * A woman at least 50 years of age with an intact uterus, not on hormone therapy, who has had either: cessation of menses for at least 1 year; or at least 6 months of spontaneous amenorrhea with a follicle stimulating hormone greater than (>)40 milli-international units per milliliter (mIU/mL); or
    * A woman 55 years or older not on hormone therapy, who has had at least 6 months of spontaneous amenorrhea; or
    * A woman at least 55 years of age with a diagnosis of menopause prior to staring hormone replacement therapy

Exclusion Criteria:

* Currently enrolled in any other clinical trial involving a study drug or device, or any other type of medical research judged not compatible with this study (Participants in the previous PRCL study (SMAD) will be allowed to be included in this study, provided that they meet all inclusion and none of the exclusion criteria)
* Participated in a clinical study within last 30 days
* Present with pustular, erythrodermic psoriasis, generalized pustular psoriasis, or acute guttate psoriasis
* Have current serious or unstable illnesses including hepatic, renal, gastroenterologic, respiratory, cardiovascular (including a history of ischemic or structural heart disease, conduction system disease or history of clinically significant arrhythmia), endocrinologic, neurologic, psychiatric, immunologic, hematologic, or dermatologic disease
* Have a history of clinically significant severe drug allergies or severe post treatment hypersensitivity reactions
* Have received inactivated vaccine within 4 weeks prior to dosing in this study, or a live vaccine within the last 3 months
* A history of clinically significant opportunistic infection (for example, invasive candidiasis or Pneumocystis pneumonia)
* Had symptomatic herpes zoster within last 3 months or other recent or ongoing infection
* Present with any of the following laboratory test results:

  * Positive QuantiFERON®-tuberculosis test
  * For women, positive serum pregnancy test
  * Evidence of Human Immunodeficiency Virus (HIV) infection or are positive for HIV antibodies
  * Positive test for active hepatitis B
  * Positive of anti-hepatitis C antibody with confirmed presence of hepatitis C virus, or chronic liver disease
* Evidence of clinically significant hepatic or renal impairment
* Clinically significant ECG (electrocardiogram) abnormalities or personal or family history of heart disease, including:

  * Confirmed corrected QT interval with Frederica's correction (QTcF) >450 milliseconds (msec) for both men and women
  * Specific bundle branch blocks, irregular rhythms, history of unexplained syncope, or family history of unexplained death
* Are receiving any of the following therapies for psoriasis:

  * Systemic retinoids within last 12 weeks
  * Systemic psoriasis therapy, such as psoralen and ultraviolet A (PUVA) light therapy, cyclosporine, corticosteroids, methotrexate, oral retinoids, mycophenolate mofetil, thioguanine, hydroxyurea, sirolimus, azathioprine, or phototherapy (including ultraviolet B or self-treatment with tanning beds or therapeutic sunbathing) within last 4 weeks
  * Topical psoriasis treatment within last 2 weeks; or
  * Any biologic agent within the following washout periods: 30 days for anti-tumor necrosis factor (TNF) inhibitors, and 90 days for other agents

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2018-09-25 (Actual); Primary Completion 2019-04-29 (Actual); Study Completion 2019-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — PRCL Research Inc.
Locations (16):
- Canada (7):
  - Wiseman Dermatology Research Inc., Winnipeg, Manitoba
  - SimcoDerm Medical and Surgical Dermatology, Barrie, Ontario
  - DermEffects, London, Ontario
  - Lynderm Research Inc., Markham, Ontario
  - SKiN Centre for Dermatology, Peterborough, Ontario
  - K. Papp Clinical Research, Waterloo, Ontario
  - Carey-Wang - Dermatology & Dermatologic Surgery Center, Westmount, Quebec
- Slovakia (6):
  - Maxderm Dermatovenerologická ambulancia, Bardejov
  - SKINKLINIK Dermatovenerologická ambulancia, Bratislava
  - BeneDerma, Bratislava
  - Derma therapy, spol., Bratislava
  - AHS Dermatology, Nitra
  - SANARE - Dermatovenerologická ambulancia, Svidník
- Ukraine (3):
  - Oleksandrivska Clinical Hospital, Department of Dermatology and Venereology, Kiev
  - LLC MK BLAGOMED, Department of Dermatology, Kyiv
  - Zaporizhzhya Regional Dermatovenereology Clinical Hospital, Zaporizhzhya

RESULTS

PARTICIPANT FLOW:
Groups:
- PRCL-02 25 Milligrams (mg): Loading dose of 150 mg followed by a once daily maintenance dose commencing on Day 2 and continuing for 12 weeks
  PRCL-02: Oral tablets
- PRCL-02 50 mg: Loading dose of 300 mg followed by a once daily maintenance dose commencing on Day 2 and continuing for 12 weeks
  PRCL-02: Oral tablets
Period: Overall Study
Arm/Group | PRCL-02 25 Milligrams (mg) | PRCL-02 50 mg | Placebo
Started | 31 | 30 | 31
Completed | 28 | 23 | 26
Not Completed | 3 | 7 | 5
Not completed — Withdrawal by Subject | 2 | 2 | 3
Not completed — Participant Did Not Return for Visit | 0 | 1 | 0
Not completed — High Neutrophils | 0 | 0 | 2
Not completed — Patient Did Not Meet Eligibility | 1 | 0 | 0
Not completed — Exacerbation of Psoriasis | 0 | 1 | 0
Not completed — Adverse Event | 0 | 2 | 0
Not completed — Dizziness and Rash | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety population
Groups:
- Total: Total of all reporting groups
Arm/Group | PRCL-02 25 Milligrams (mg) | PRCL-02 50 mg | Placebo | Total
Number analyzed (Participants) | 31 | 30 | 31 | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 30 | 29 | 29 | 88
  >=65 years | 1 | 1 | 2 | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 8 | 33
  Male | 17 | 19 | 23 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 31 | 30 | 31 | 92
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 27 | 29 | 31 | 87
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 0 | 2
Region of Enrollment [Number; unit: participants]
  Canada | 9 | 7 | 6 | 22
  Ukraine | 9 | 10 | 15 | 34
  Slovakia | 13 | 13 | 10 | 36

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Psoriasis Area and Severity Index ≥75% (PASI 75) Improvement
Description: Following 12 weeks of treatment. The Psoriasis Area and Severity Index (PASI) scores the severity of disease on a scale from 0 to 72 (where a score of 72 indicates extreme disease severity). PASI 75 indicates 75% improvement from baseline to Week 12 in the Psoriasis Area and Severity Index
Time Frame: Baseline to week 12
Population: Intent to treat population
Measure: Count of Participants; unit: Participants
Arm/Group | PRCL-02 25 Milligrams (mg) | PRCL-02 50 mg | Placebo
Number analyzed (Participants) | 30 | 29 | 31
Participants | 4 | 1 | 0

2. Secondary Outcome: Number of Participants With Any Treatment Emergent Adverse Event
Description: Following 12 weeks of treatment
Time Frame: Baseline up to week 18
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | PRCL-02 25 Milligrams (mg) | PRCL-02 50 mg | Placebo
Number analyzed (Participants) | 31 | 30 | 31
Participants | 14 | 12 | 10

3. Secondary Outcome: Area Under the Concentration Time Curve (AUC0-τ)
Description: Steady state after 12 weeks of treatment
Time Frame: Predose and 1, 2, 4, 8, 336, 672, 1008, 1344 hours post dose, on Day 84
Population: Pharmacokinetic (PK) evaluable
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*mg/mL
Arm/Group | PRCL-02 25 Milligrams (mg) | PRCL-02 50 mg
Number analyzed (Participants) | 24 | 20
h*mg/mL | 165000 (627) | 439000 (492)

4. Secondary Outcome: Maximum Observed Drug Concentration (Cmax)
Description: Steady state after 12 weeks of treatment
Time Frame: Predose and 1, 2, 4, 8, 336, 672, 1008, 1344 hours post dose, on Day 84
Population: Pharmacokinetic (PK) evaluable
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PRCL-02 25 Milligrams (mg) | PRCL-02 50 mg
Number analyzed (Participants) | 24 | 20
ng/mL | 984 (200) | 2220 (139)

5. Secondary Outcome: Time to Reach Maximum Observed Drug Concentration (Tmax)
Description: Steady state after 12 weeks of treatment
Time Frame: Predose and 1, 2, 4, 8, 336, 672, 1008, 1344 hours post dose, on Day 84
Population: Pharmacokinetic (PK) evaluable
Measure: Median (Full Range); unit: hours
Arm/Group | PRCL-02 25 Milligrams (mg) | PRCL-02 50 mg
Number analyzed (Participants) | 24 | 20
hours | 2.0 [0 to 8.12] | 4.00 [0 to 358]

ADVERSE EVENTS:
Time Frame: 20 weeks
Arm/Group | PRCL-02 25 Milligrams (mg) | PRCL-02 50 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/30 | 0/31
Serious Adverse Events (participants affected / at risk) | 1/31 | 0/30 | 0/31
Other Adverse Events (participants affected / at risk) | 3/31 | 3/30 | 4/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PRCL-02 25 Milligrams (mg) (N=31) | PRCL-02 50 mg (N=30) | Placebo (N=31)
Measles (Infections and infestations) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PRCL-02 25 Milligrams (mg) (N=31) | PRCL-02 50 mg (N=30) | Placebo (N=31)
Nausea (Gastrointestinal disorders) | 1 | 2 | 0
Psoriatic arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Recurrent psoriatic arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2
Dizziness (Nervous system disorders) | 2 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-07-20): https://cdn.clinicaltrials.gov/large-docs/78/NCT03614078/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-03): https://cdn.clinicaltrials.gov/large-docs/78/NCT03614078/SAP_001.pdf